CLINICAL TRIAL: NCT02315183
Title: An Observational Case Control Study to Identify the Role of MV and MV Derived Micro-RNA in Post CArdiac Surgery Acute Kidney Injury: The MaRACAS Study
Brief Title: An Observational Case Control Study to Identify the Role of MV and MV Derived Micro-RNA in Post CArdiac Surgery AKI
Acronym: MaRACAS
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0419
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2014-12

CONDITIONS: Acute Kidney Injury
Keywords: Post cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine samples are taken at numerous timepoints upto 5 days post cardiac surgery.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: This is an observational Study — THis study has no intervention
  Other Names: MaRACAS Study

SUMMARY:
Acute kidney injury (AKI) complicates over 25% of cardiac surgical procedures where it increases mortality up to fourfold. The incidence of AKI is increasing, the pathogenesis is poorly understood, current diagnostic tests lack specificity and sensitivity, and there is no effective treatment. Improving outcomes in patients at risk of AKI has recently been defined as an NHS priority. The primary aim of this study is to determine how plasma derived microvesicles (MV) or more specifically MV associated microRNAs (miRNA) regulate survival and signalling in post cardiac surgery AKI. The study involves a clinical and experimental research project that will combine laboratory analyses of circulating MV and miRNA from clinical studies. The study will specifically consider how MV and miRNA alter inflammatory signaling in kidneys after cardiac surgery, how these are modified by important clinical risk factors, and whether they may serve as early biomarkers of injury.

DETAILED DESCRIPTION:
AKI is characterised by upregulation of competing pro-survival and pro- inflammatory/ apoptotic signaling pathways whereby processes associated with renal recovery; tubular epithelial phenotypic change and proliferation occur simultaneously with those associated with diminished GFR, vascular inflammation, tubular dysfunction and epithelial apoptosis. Protection from AKI can be achieved by altering the balance of these pathways; for example upregulation of the pivotal phosphatidylinositol 3-kinase - serine-threonine protein kinase B (PI3K-Akt) pro-survival pathway following the administration of erythropoietin or insulin like growth factor inhibits experimental AKI following renal ischaemia and reperfusion in rodents and swine. In our own work we have shown that post cardiopulmonary bypass (CPB) AKI in swine can be prevented by the administration of either a phosphodiesterase type 5 (PDE-5) inhibitor which promotes cell survival and endothelial homeostasis via augmentation of endogenous nitric oxide (NO) signalling, or by the inhibition of endothelin-1 (ET-1), an important pro-inflammatory mediator and promoter of oxidative stress in renal injury How these competing pathways are regulated in patients at risk of AKI is poorly understood however, and it is our belief that the identification of these processes will facilitate the development of new and effective prevention and treatment strategies for AKI and improved outcomes for patients

ELIGIBILITY:
Inclusion Criteria:

1. Adult cardiac surgery patients (>16 years) undergoing coronary artery bypass grafting or valve surgery with moderately hypothermic CPB (32-34°C) blood cardioplegia.
2. Identified as being at increased risk for AKI from a modified risk score.

Exclusion Criteria:

1. Patients with pre-existing inflammatory state: sepsis undergoing treatment, acute kidney injury within 5 days, chronic inflammatory disease, congestive heart failure,
2. Emergency or salvage procedure,
3. Ejection fraction <30 %,
4. Patient in a critical preoperative state (Kidney Disease: Improving Global Outcomes (KDIGO) Stage 3 AKI or requiring ionotropes, ventilation or intra-aortic balloon pump).
5. Pregnancy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be carried out at a large tertiary academic cardiac surgery unit in the UK; the University Hospitals of Leicester NHS Trust. This unit performs over 1,200 major cardiac procedures per year, of which 300 are expected to develop acute kidney injury.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
AKI defined according to the KDIGO criteria or by urine NGAL levels >150nmol/mg at 6 hours postoperatively. | 2 Years

SECONDARY OUTCOMES:
Data on demographics, perioperative clinical characteristics and medications. | 2 Years
MV will be isolated from arterial blood samples collected prior to anaesthetic induction, at chest closure and at 6 and 24 hours postoperatively, and characterised using flow cytometry and NanoSight LM10 (Nanosight, London, UK). | 2 Years
Likely sources of MV will also be evaluated; Platelet and monocyte activation and aggregation will be determined by flow cytometry, endothelial activation will be determined by ELISA measurement of circulating ICAM and E-selectin in serum. | 2 Years
MV associated miRNA profiles will be determined using microarray in patients with AKI (n=6 diabetic, n=6 non diabetic) and a matched control group (n=6 diabetic, n=6 non diabetic) without AKI. | 2 Years
The systemic inflammatory response will be quantified by measurement of serum IL-8 and IL-6. | 2 Years
Renal inflammation will be determined by urine Neutrophil Gelatinase-Associated Lipocalin (NGAL) and Liver type- Fatty Acid Binding Protein (L-FABP) measured at baseline, and then at 6 and 24 hours postoperatively. | 2 Years
MV and MV associated miRNA signaling will be evaluated ex vivo in a micro fluidics model. | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Murphy, Prof, Principal Investigator — University of Leicester
Locations (1):
- Department of Cardiovascular Sciences., Leicester, Leicestershire, United Kingdom